CLINICAL TRIAL: NCT03653130
Title: Participatory Music Program for Homeless Veterans (Crossroads Orchestra): Pilot Evaluation
Brief Title: Participatory Music Program for Homeless Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Quality Enhancement Research Intiative (Other)
Responsible Party: Principal Investigator, Dawn M. Bravata, Professor of Medicine and Adjunct Professor of Neurology, VA Quality Enhancement Research Intiative
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1802361597
Record Dates: First submitted 2018-08-21; First posted 2018-08-31 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Quality of Life
Keywords: homeless; recreational therapy; community integration; reintegration; Veteran; housing insecurity; Domiciliary; Human Occupation; Occupational therapy; Music

STUDY DESIGN:
Intervention Model Description: Parallel Interventional Study Model: Intervention participants (N=40) and usual care controls (N=40) will be eligible if they are residents of the Indianapolis VA Domiciliary who are eligible to participate in elective activities at the time of recruitment. Intervention participants will include eligible Veterans who agree to participate in the intervention. Usual Care Controls will include eligible Veterans who agree to complete the interviews and measures, but do not agree to participate in the participatory music program. Records for retrospective chart review (N=160) will be selected from past Domiciliary residents based on case-matching for gender and biological sex factors with intervention participants.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Program (Experimental): Participants will receive an instrument (violin, viola, or cello). Intervention sessions will take place twice a week at the Domiciliary and once per week at the Domiciliary or at a community location (Richard L. Roudebush VA Medical Center or Regenstrief Institute). Each session will include: thirty minutes of group music instruction by an experienced music educator with skills in adult music education followed by thirty minutes of weekly adult ensemble experience.
  Interventions: Behavioral: Crossroads Orchestra Participatory Music Program
- Usual Care Control (No Intervention): Usual care at VA Domiciliary including participation in Domiciliary recreational therapy electives (if eligible).
- Retrospective Chart Review (No Intervention): Retrospective chart reviews case-matched to intervention participants for age and biological sex factors.

INTERVENTIONS:
Behavioral: Crossroads Orchestra Participatory Music Program — The intervention is a participatory music program where adults engage in music-making as members of a strings orchestra.
  Arms: Intervention Program

SUMMARY:
This pilot project evaluates the effectiveness of a participatory music program for Veterans cared for in the Domiciliary Care for Homeless Veterans (DCHV) Program (Indianapolis, IN) in terms of improving quality of life. A secondary goal of this study is to evaluate the effect of the participatory music program on community reintegration and healthcare utilization. The participatory music program entitled the "Crossroads Orchestra" includes both music education and an orchestra experience. The objective of this intervention program is to use an engaging music-based education and group orchestra experience to provide participants with an avocation that will improve their quality of life and facilitate their reintegration into the community. The Crossroads Orchestra pilot project protocol has been grounded on concepts from occupational therapy and recreational therapy; specifically, providing participants with a meaningful new activity that is enjoyable, that can be provided across a spectrum of skill levels (e.g., for participants with no musical training as well as for individuals who are proficient strings musicians), and that can provide participants with a new sense of self.

DETAILED DESCRIPTION:
SPECIFIC AIMS:

Aim 1: To evaluate the effectiveness of the participatory music program in terms of improving quality of life.

Aim 2: To evaluate the effect of the participatory music program on community reintegration. Veteran members of the Crossroads Orchestra program may develop a sense of participating in something that "is bigger than oneself." They may develop a new sense of self, or identify with a new role. They may develop a sense of commitment to their stand-partner. These positive new perspectives may facilitate their transition from the Domiciliary to the community. Semi-structured interviews with participants will be conducted to understand participants' experiences to both improve the program and to assess its effects. The Military to Civilian Questionnaire (M2C-Q) measure will be used to assess community reintegration.

Secondary Aim: To evaluate the effect of the participatory music program on healthcare utilization. This pilot project is not powered to identify statistically significant differences in healthcare utilization but rather is designed to provide preliminary data to understand the potential role of a music education and orchestra participation experience for improving outcomes among Veteran participants.

INTERVENTION DESCRIPTION:

The intervention is a participatory music program where adults engage in music-making as members of a strings orchestra. As part of the Crossroads Orchestra, participants will receive an instrument (violin, viola, or cello). The intervention sessions will take place twice a week at the Domiciliary and once per week at either the Domiciliary or other Indianapolis community location. Each session will include: thirty minutes of group music instruction by an experienced music educator with skills in adult music education followed by thirty minutes of weekly adult ensemble experience. The choice of music pieces will be made by the interventionist in consultation with participants (to ensure that the choices represent selections that are most engaging for the majority of participants). The participants will be given a binder with sheet music and practice logs. The music educator will create Youtube videos demonstrating violin, viola, and cello techniques and providing helpful tips. Participants will be encouraged to practice and to attend all of the group sessions.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the Indianapolis VA Domiciliary who are eligible to participate in elective activities (i.e., they have been Domiciliary residents for a minimum of two weeks and they have not committed any infractions that would place them on restriction status)

Exclusion Criteria:

* Visual impairment (blindness)
* Profound hearing impairment (deafness)
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Quality of Life: 20-Item Short Form Health Survey (SF-20) | change from baseline to month-6
  We will examine the trajectory of quality of life scores over time utilizing the SF-20. The total score ranges from 0-100, higher values indicate better functioning.

SECONDARY OUTCOMES:
Community Reintegration: Military to Civilian Questionnaire (M2C-Q) | 1 month post-transition
  We will use the M2C-Q measure to assess perceived difficulties reintegrating into community life after leaving the Domiciliary. This is a 16 item scale where each item is scored on a 5-point Likert scale with 0 representing no difficulty and 4 representing extreme difficulty with reintegration.

OTHER OUTCOMES:
Healthcare Utilization: Chart Review | One-year pre-enrollment versus the one-year post-enrollment period
  Healthcare utilization includes ED visits, inpatient admissions, and clinic missed appointments ("no shows")
Flow State (Experience of Total Absorption): Flow State Scale (FSS-2) | month-6
  Flow state describes a participant's engagement with the intervention. The FSS-2 includes 9 items that are scored from 1 (disagree) to 5 (strongly agree). Higher scores indicate a greater degree of task absorption.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Bravata, MD, Principal Investigator — VA Quality Enhancement Research Initiative
Locations (1):
- VA Domiciliary, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Keiper S, Sandene, B.A., Persky, H.R., and Kuang, M. . The Nation's Report Card: Arts 2008 Music & Visual Arts (NCES 2009-488). In: National Center for Education Statistics IoES, U.S. Department of Education, ed. Washington, D.C.2009. — https://files.eric.ed.gov/fulltext/ED505664.pdf
- See also: Ending Veteran Homelessness: A Community by Community Tally — https://www.va.gov/homeless/endingvetshomelessness.asp